CLINICAL TRIAL: NCT02859103
Title: A Dimensional Approach to Evaluate Reward Processing in Major Depressive Disorder Before and After Treatment With Desvenlafaxine
Brief Title: Dimensional Approach to Evaluate Reward Processing in Major Depressive Disorder Pre- and Post-Desvenlafaxine Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Sakina Rizvi, Scientist, Unity Health Toronto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DVS-01
Record Dates: First submitted 2016-07-15; First posted 2016-08-08 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Depression; Anhedonia
MeSH Terms: conditions — Depression; Anhedonia | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Patients in this arm will receive treatment with desvenlafaxine for 8 weeks.
  Interventions: Drug: Desvenlafaxine
- Healthy Control (No Intervention): Patients in this arm are healthy controls and will not receive any medication.

INTERVENTIONS:
Drug: Desvenlafaxine — Patients will be provided 50mg dose of desvenlafaxine for 1 week titrated up to 100mg dose of desvenlafaxine for 7 weeks.
  Other Names: Pristiq
  Arms: Treatment

SUMMARY:
Anhedonia (the lack of pleasure in normally pleasurable things) is a common symptom of major depressive disorder (MDD), and it may impact how patients with depression experience reward. Understanding how anhedonia is related to the experience of reward may help improve how depression is treated. Computer tasks can be used to measure how reward is experienced, and these measures might be able to predict things like who is likely to become depressed, or who will respond to antidepressant medication. Studying the relationship between anhedonia and reward in patients with depression might also tell us something about how to improve diagnosis and treatment of other psychiatric disorders.This is an open label controlled treatment study lasting 8 weeks. The brain scans will be used to find changes in brain areas that may be related to how people perform on the tasks. The investigators goal is to use this information to help us find a reliable predictor that can be used to guide MDD treatment.

ELIGIBILITY:
Inclusion/exclusion criteria for MDD patients (n=40) are as follows:

Inclusion Criteria

1. DSM-5 criteria for Major Depressive Episode (MDE) within a MDD, confirmed through MINI diagnosis
2. Age between 18 and 60 years
3. Hamilton Depression Rating Scale - 17 item (HRSD-17)58 > 17 (moderate to severe symptoms)
4. Free of psychotropic medications for at least 5 half-lives before baseline visit
5. Ability to undergo MRI scanning (absence of metal, pacemakers, etc.)

Exclusion Criteria

1. Pregnancy/lactation
2. Medical condition requiring immediate investigation or treatment
3. Recent (< 6 months)/current history of drug abuse/dependence (other than caffeine, or nicotine)
4. Lifetime history of psychosis, other Axis I comorbidities are allowable
5. Significant Axis II diagnosis
6. Previous intolerance or failure to respond to an adequate trial of desvenlafaxine
7. Failure of > 2 antidepressant treatments of adequate dose and duration for current MDE

Inclusion/exclusion criteria for Healthy Controls (n=20) are as follows:

Inclusion Criteria

1. Age between 18 and 60 years
2. Ability to undergo MRI scanning (absence of metal, pacemakers, etc.)

Exclusion Criteria

1. Pregnancy/lactation
2. Medical condition requiring immediate investigation or treatment
3. Lifetime history of any psychiatric disorder
4. Lifetime history of receiving an antidepressant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Measuring Reward association and valuation using the Reward Association Task | Change from Baseline at 8 Weeks
  Based on signal detection theory, it evaluates response bias as a function of prior reward and permits an objective assessment of disorder-related sensitivity to reward. To evaluate the how the 6 facets of reward are related to each other in unmedicated MDD patients in order to develop a clearer understanding of reward pathways
Measuring Expectation using a prediction error task, to measure learning and choosing, during functional Magnetic Resonance Imaging (fMRI) | Change from Baseline at 8 Weeks
  This distinction was included in the design in order to dissociate potentially different neural circuits subserving learning reward associations and using them to guide behavior. To evaluate the how the 6 facets of reward are related to each other in unmedicated MDD patients in order to develop a clearer understanding of reward pathways
Anticipation of reward using the monetary incentive delay during fMRI | Change from Baseline at 8 Weeks
  This task was designed to disentangle anticipatory vs. consummatory phases of reward processing. To evaluate the how the 6 facets of reward are related to each other in unmedicated MDD patients in order to develop a clearer understanding of reward pathways
Motivation/effort using the Cued-Reinforcement Reaction Time Task and the EEfRT task. | Change from Baseline at 8 Weeks
  The Cued-Reinforcement Reaction Time Task (CRRT) provides an evaluation of reward-based reaction time speed as an index of incentive motivation.The EEfRT task allows analysis of the predictive value of reward probability and magnitude on effort-based decision making. To evaluate the how the 6 facets of reward are related to each other in unmedicated MDD patients in order to develop a clearer understanding of reward pathways
Pleasure/Liking using the monetary incentive delay task in an fMRI | Change from Baseline at 8 Weeks
  This task was designed to disentangle anticipatory vs. consummatory phases of reward processing. To evaluate the how the 6 facets of reward are related to each other in unmedicated MDD patients in order to develop a clearer understanding of reward pathways. To evaluate the how the 6 facets of reward are related to each other in unmedicated MDD patients in order to develop a clearer understanding of reward pathways
Feedback integration using the Probabilistic Reversal Learning task during fMRI | Change from Baseline at 8 Weeks
  participants are presented with a choice of two stimuli. Based on their first choice, the selected stimulus will be rewarded with a high probability, while the other will be rewarded with a low probability.To evaluate the how the 6 facets of reward are related to each other in unmedicated MDD patients in order to develop a clearer understanding of reward pathways

CONTACTS AND LOCATIONS:
Overall Officials: Sakina Rizvi, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No